CLINICAL TRIAL: NCT00457366
Title: A Comparison Study of the Efficacy of a Rapid Titration of Quetiapine and Haloperidol in Agitated Adults in an Emergency Setting.
Brief Title: A Comparison Study of the Efficacy of Quetiapine and Haloperidol in Agitated Adults in Emergency Room
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-05-00331
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2017-04

CONDITIONS: Agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Quetiapine Fumarate; Haloperidol; Lorazepam; Benztropine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Quetiapine (Active Comparator): Quetiapine is being used in an ER setting on agitated patients, being administered orally.
  Interventions: Drug: Quetiapine
- Haloperidol (Active Comparator): "Haloperidol" is being used in an ER setting on agitated patients, administered IM. This is being used in combination with lorazepam and cogentin. We are comparing the use of this "cocktail" to quetiapine alone.
  Interventions: Drug: Haloperidol
- Lorazepam (Active Comparator): "Lorazepam" is being used in an ER setting on agitated patients, administered IM.This is being used in combination with haloperidol, and cogentin. We are comparing the use of this "cocktail" to quetiapine alone.
  Interventions: Drug: Lorazepam
- Cogentin (Active Comparator): "Cogentin" is being used in an ER setting on agitated patients, administered IM.
  This is being used in combination with haloperidol, and lorazepam. We are comparing the use of this "cocktail" to quetiapine alone.
  Interventions: Drug: Cogentin

INTERVENTIONS:
Drug: Quetiapine — Quetiapine 300mg PO/Initial dose and repeat dose at 2 hours if deemed clinically necessary up to a maximum dose of Quetiapine 600mg PO QD
  Other Names: no other name
  Arms: Quetiapine
Drug: Haloperidol — given in combination with Lorazepam 2 mg IM, Cogentin 2 mg IM; repeated at 2 hours as deemed clinically necessary
  Other Names: no other names
  Arms: Haloperidol
Drug: Lorazepam — given in combination with Haloperidol 5mg IM and cogentin 2mg IM; repeated at 2 hours as deemed clinically necessary.
  Other Names: no other name
  Arms: Lorazepam
Drug: Cogentin — given in combination with haloperidol 5mg IM, and Lorazepam 2mg IM; repeated at 2 hours as deemed clinically necessary.
  Other Names: no other name
  Arms: Cogentin

SUMMARY:
In the Psychiatric Emergency Room, agitated patients are treated routinely with an I.M. Haloperidol "cocktail" (Haloperidol 5 mg, Lorazepam 2 mg, Cogentin 2 mg), which has proved to be an effective treatment. However, since it is an intramuscular injection, it is more complicated and perhaps less acceptable to patients as well as more likely to cause EPS (extrapyramidal symptoms). Of late in our emergency room, we started using high dose Quetiapine 300 mg PO to replace the "cocktail" for treating agitation. It has shown promising results.

DETAILED DESCRIPTION:
In the Psychiatric Emergency Room, agitated patients are treated routinely with an I.M. Haloperidol "cocktail" (Haloperidol 5 mg, Lorazepam 2 mg, Cogentin 2 mg), which has proved to be an effective treatment. However, since it is an intramuscular injection, it is more complicated and perhaps less acceptable to patients as well as more likely to cause EPS (extrapyramidal symptoms). Of late in our emergency room, we started using high dose Quetiapine 300 mg PO to replace the "cocktail" for treating agitation. It has shown promising results.

This study is designed to compare the efficacy and safety of Quetiapine with the routine "cocktail for treatment of agitation.

The primary purpose of this study is to determine the efficacy and safety of Quetiapine by using high dose Quetiapine (300 mg) PO to treat agitated patients in the psychiatric emergency room.

The secondary purpose is to test the immediate effect on agitation caused by illicit drug abuse or the alcohol abuse.

ELIGIBILITY:
Inclusion Criteria:

1. English or Spanish speaking patients
2. Provision of written informed consent-English and Spanish
3. Males and females age 18 to 60 years. Females who are pregnant by inspection should not be included.
4. Provision at diagnosis meeting the Diagnostic and Statistical Manual of Mental Disorder, 4th edition (DSM-IV) criteria for Axis I documented who present in an agitated state. PANSS-EC score should be >15.
5. Ability, in the treating physician's opinion, to co-operate with taking oral medication

Exclusion Criteria:

1. Pregnant females who will thus receive routine care in the treating physician's opinion
2. Unstable medical illness
3. Withdrawal stage from any illicit drugs
4. Psychosis that prohibits participation in trial
5. Females of childbearing age where pregnancy cannot be confirmed or denied by screening
6. Patients who required continued intervention or prolonged restraint

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George M Simpson, MD, Principal Investigator — USC+LAC Medical Center
Locations (1):
- Los Angeles County Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Quetiapine: Quetiapine is being compared to a "cocktail" consisting of haloperidol, lorazepam, and cogentin to see which works best in agitated patients that are being brought into the ER.
- "Cocktail" Consisting of Haloperidol, Lorazepam, Cogentin: This "cocktail" consisting of haloperidol, lorazepam, and cogentin is being compared to quetiapiene to see which works best in agitated patients that are being brought into the ER.
Period: Overall Study
Arm/Group | Quetiapine | "Cocktail" Consisting of Haloperidol, Lorazepam, Cogentin
Started | 40 | 32
Completed | 40 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 72 patients were included in the study. 4 patients were randomized to the Haloperidol cocktail group but were excluded from the analysis because they only had demographic data. Analyses were performed on the resulting 68 patients who had clinical outcome data available.
Groups:
- Quetiapine: Quetiapine
  Quetiapine: Quetiapine 300mg PO/Initial dose and repeat dose at 2 hours if deemed clinically necessary upto a maximum dose of Quetiapine 600mg PO QD
- Cocktail: Cocktail (Haloperidol, Lorazepam, Cogentin)
  Cocktail (Haloperidol, Lorazepam, Cogentin): Haloperidol 5 mg im, Lorazepam 2 mg im, Cogentin 2 mg im; repeated at 2 hours as deemed clinically necessary
- Total: Total of all reporting groups
Arm/Group | Quetiapine | Cocktail | Total
Number analyzed (Participants) | 38 | 34 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 34 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 36.1 [18 to 60] | 35.8 [18 to 60] | 36.0 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 29 | 28 | 57
Region of Enrollment [Number; unit: participants]
  United States | 38 | 34 | 72

OUTCOME MEASURES:

1. Primary Outcome: Change in the PANSS-EC Score Among Participants From Baseline to 2 Hours After Administration of the Medication.
Description: The PANSS-EC is the Positive and Negative Syndrome Score - Excited Component, which includes 5 items (excitement, hostility, tension, uncooperative, poor impulse control), which are rated from 1 (not present) to 7 (extremely severe); scores range from 5 to 35; mean scores ≥ 20 clinically correspond to severe agitation. This set of items detects differences between drug and placebo when evaluating acute agitation and aggression in psychiatric patients with different psychiatric pathologies (Montoya, A; Villadares, A; Lizan, L, et al., 2011).
Time Frame: Two hours
Population: 34 patients received the Cocktail, but 4 of these were excluded from the analysis because they had only demographic data and no clinical outcome data. A total of 38 patients received Quetiapine; all were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Cocktail: Cocktail (Haloperidol, Lorazepam, Cogentin): Haloperidol 5 mg im, Lorazepam 2 mg im, Cogentin 2 mg im; repeated at 2 hours as deemed clinically necessary.
- Quetiapine: Quetiapine 300 mg PO
Arm/Group | Cocktail | Quetiapine
Number analyzed (Participants) | 30 | 38
score on a scale | -11.0 (0.82) | -11.5 (0.69)
Statistical Analysis 1: Comparison: Cocktail vs Quetiapine; Test type: Other — We used an analysis of covariance (ANCOVA) with baseline as the covariate to analyze the PANSS-EC at hour 2; p > 0.05, ANCOVA

ADVERSE EVENTS:
Arm/Group | Quetiapine | Cocktail
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/32
Other Adverse Events (participants affected / at risk) | 0/40 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No